CLINICAL TRIAL: NCT01449669
Title: Skeletal Muscle and Plasma Concentrations of Cefazolin During Pediatric Cardiac Surgery Utilizing Cardiopulmonary Bypass, Deep Hypothermic Cardiac Arrest, and Modified Ultrafiltration
Brief Title: Surgical Site Infection Study
Acronym: SSI
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 11-007976; PSSIMD
Record Dates: First submitted 2011-09-26; First posted 2011-10-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Cava-pulmonary Anastomosis
Keywords: pharmacokinetics; cefazolin; microdialysis sampling; interstitial fluid; skeletal muscle; plasma; children

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of cefazolin using both plasma and microdialysate sampling methods in children with single ventricle physiology undergoing their second palliation procedure. This will provide data to determine if the current standard dosing regimen of cefazolin is adequate to achieve and maintain tissue concentrations greater than the minimum inhibitory concentrations (MIC) for common post-surgical pathogens that cause Surgical Site Infections (SSIs).

DETAILED DESCRIPTION:
This study aims to sample interstitial fluid (IF) of infants undergoing superior cava-pulmonary anastomosis (either Glenn or Hemi-Fontan) cardiac surgical procedures who receive cefazolin as their surgical prophylactic antibiotic. Cefazolin concentrations will then be determined in both microdialysate and plasma samples and used to define the pharmacokinetics of cefazolin at the tissue level and compare that to plasma pharmacokinetics. In addition, the data gathered will be used to assess how cardiopulmonary bypass (CPB), deep hypothermic cardiac arrest (DHCA), and modified ultrafiltration (MUF) affect tissue penetration of the prophylactically administered cefazolin.

The study involves the use of microdialysis (MD) and plasma sampling methods to determine the pharmacokinetic properties of cefazolin when used as a prophylactic antibiotic during the second palliation procedure (superior vena cava-pulmonary anastomosis) for infants with single ventricle physiology. This requires the use of microdialysis (MD) catheters inserted into the left deltoid muscle in eligible subjects after the induction of general anesthesia as well as collection of microdialysate and blood samples throughout the duration of the procedure. Cefazolin will be administered as standard of care. Cefazolin concentrations in the collected samples will be measured via a validated high-performance liquid chromatography (HPLC) and mass spectrometry assay. Pharmacokinetic analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with single ventricle physiology undergoing their second palliation procedure (typically performed between 3-6 months of age)
* Use of cefazolin as the prophylactic antibiotic during the operation
* Written informed consent provided by the parent or legal guardian

Exclusion Criteria:

* Use of prophylactic antibiotic other than cefazolin during the operation
* Anatomic or other abnormalities of the upper arm that would preclude insertion of a microdialysis catheter
* Known renal or hepatic function

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Males or females with single ventricle physiology undergoing their second palliation procedure (typically performed between 3-6 months of age)
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Cefazolin | predose, .08,.25, .5, 1, 1.5, 2, 3, 4 hours and post dose.
  Composite (or Profile) of Pharmacokinetics

SECONDARY OUTCOMES:
Investigate the relationship between cefazolin concentrations in the plasma and those at the level of IF of skeletal muscle | One Year
  * Investigate the effects of CPB, DHCA, and MUF on tissue distribution of cefazolin
  * Determine the concentration of cefazolin in IF of skeletal muscle at different stages of cardiac surgery and compare these values to concentrations of cefazolin needed to be effective against common bacterial organisms causing SSIs
  * Investigate the relationship between cefazolin concentrations in the plasma and those at the level of IF of skeletal muscle.
  * Assess the safety of the use of microdialysis method during pediatric cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Todd Kilbaugh, MD, Principal Investigator — Children's Hospital of Philadelphia

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Division of Healthcare Quality Promotion (DHPQ). Estimates of Healthcare-Associated Infections. March 12, 2010. Available at: http://www.cdc.gov/ncidod/dhqp/hai.html. Accessed August 3, 2010.
- [Background] Anderson DJ, Kaye KS, Classen D, Arias KM, Podgorny K, Burstin H, Calfee DP, Coffin SE, Dubberke ER, Fraser V, Gerding DN, Griffin FA, Gross P, Klompas M, Lo E, Marschall J, Mermel LA, Nicolle L, Pegues DA, Perl TM, Saint S, Salgado CD, Weinstein RA, Wise R, Yokoe DS. Strategies to prevent surgical site infections in acute care hospitals. Infect Control Hosp Epidemiol. 2008 Oct;29 Suppl 1:S51-61. doi: 10.1086/591064. No abstract available. PMID 18840089
- [Background] Sparling KW, Ryckman FC, Schoettker PJ, Byczkowski TL, Helpling A, Mandel K, Panchanathan A, Kotagal UR. Financial impact of failing to prevent surgical site infections. Qual Manag Health Care. 2007 Jul-Sep;16(3):219-25. doi: 10.1097/01.QMH.0000281058.99929.ea. PMID 17627217
- [Background] Costello JM, Graham DA, Morrow DF, Morrow J, Potter-Bynoe G, Sandora TJ, Pigula FA, Laussen PC. Risk factors for surgical site infection after cardiac surgery in children. Ann Thorac Surg. 2010 Jun;89(6):1833-41; discussion 1841-2. doi: 10.1016/j.athoracsur.2009.08.081. PMID 20494036
- [Background] Ben-Ami E, Levy I, Katz J, Dagan O, Shalit I. Risk factors for sternal wound infection in children undergoing cardiac surgery: a case-control study. J Hosp Infect. 2008 Dec;70(4):335-40. doi: 10.1016/j.jhin.2008.08.010. Epub 2008 Oct 31. PMID 18951662
- [Background] Holzmann-Pazgal G, Hopkins-Broyles D, Recktenwald A, Hohrein M, Kieffer P, Huddleston C, Anshuman S, Fraser V. Case-control study of pediatric cardiothoracic surgical site infections. Infect Control Hosp Epidemiol. 2008 Jan;29(1):76-9. doi: 10.1086/524323. PMID 18171193
- [Background] Kagen J, Lautenbach E, Bilker WB, Matro J, Bell LM, Dominguez TE, Gaynor JW, Shah SS. Risk factors for mediastinitis following median sternotomy in children. Pediatr Infect Dis J. 2007 Jul;26(7):613-8. doi: 10.1097/INF.0b013e31806166bb. PMID 17596804
- [Background] Allpress AL, Rosenthal GL, Goodrich KM, Lupinetti FM, Zerr DM. Risk factors for surgical site infections after pediatric cardiovascular surgery. Pediatr Infect Dis J. 2004 Mar;23(3):231-4. doi: 10.1097/01.inf.0000114904.21616.ba. PMID 15014298
- [Background] Nateghian A, Taylor G, Robinson JL. Risk factors for surgical site infections following open-heart surgery in a Canadian pediatric population. Am J Infect Control. 2004 Nov;32(7):397-401. doi: 10.1016/j.ajic.2004.03.004. PMID 15525914
- [Background] Mehta PA, Cunningham CK, Colella CB, Alferis G, Weiner LB. Risk factors for sternal wound and other infections in pediatric cardiac surgery patients. Pediatr Infect Dis J. 2000 Oct;19(10):1000-4. doi: 10.1097/00006454-200010000-00012. PMID 11055604